CLINICAL TRIAL: NCT01774604
Title: Rectal Indomethacin to Prevent Post-ERCP Pancreatitis
Brief Title: Rectal Indomethacin to Prevent Post-Endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CPHS#23749
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: Post ERCP acute pancreatitis; Post Fine Needle Aspiration (FNA) acute pancreatitis; Indomethacin; Rectal Non Steroidal Anti-Inflammatory Drugs (NSAIDs)
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indomethacin (Experimental): Indomethacin 100 mg Per Rectum (PR) x 1 in peri-procedural period
  Interventions: Drug: Indomethacin
- Placebo (Placebo Comparator): Placebo suppositories (#2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indomethacin — 100 mg Indomethacin PR x 1
  Arms: Indomethacin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether peri-procedural administration of rectal indomethacin, compared to placebo, can reduce the incidence of post-ERCP pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for an ERCP at Dartmouth-Hitchcock
2. Age greater than 18 years old
3. Ability to provide written informed consent

Exclusion Criteria:

1. Inability to provide written informed consent
2. ERCP being performed for diagnosis and/or treatment of acute pancreatitis
3. Current ongoing acute pancreatitis
4. Previously documented allergy to Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)
5. Contra-indication to NSAID therapy (creatinine level >1.4 or active peptic ulcer disease), already taking NSAIDs (other than aspirin therapy for cardioprotection)
6. Pregnant or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Levenick, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Levenick JM, Gordon SR, Fadden LL, Levy LC, Rockacy MJ, Hyder SM, Lacy BE, Bensen SP, Parr DD, Gardner TB. Rectal Indomethacin Does Not Prevent Post-ERCP Pancreatitis in Consecutive Patients. Gastroenterology. 2016 Apr;150(4):911-7; quiz e19. doi: 10.1053/j.gastro.2015.12.040. Epub 2016 Jan 9. PMID 26775631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients who presented to Dartmouth-Hitchcock Medical Center for Endoscopic Retrograde Cholangiopancreatography (ERCP) for any reason between March 2013 and December 2014
Groups:
- Placebo: Placebo suppositories (#2)
  Placebo
Period: Overall Study
Arm/Group | Indomethacin | Placebo
Started | 223 | 226
Completed | 223 | 226
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patient randomized to receive rectal indomethacin or placebo
Groups:
- Indomethacin: Indomethacin 100 mg PR x 1 in peri-procedural period
  Indomethacin: 100 mg Indomethacin PR x 1
- Total: Total of all reporting groups
Arm/Group | Indomethacin | Placebo | Total
Number analyzed (Participants) | 223 | 226 | 449
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (23.7) | 64.3 (15.1) | 64.6 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 118 | 236
  Male | 105 | 108 | 213
Indication [Number; unit: participants]
  Acute Cholangitis | 12 | 13 | 25
  Choledocholithiasis | 59 | 52 | 111
  Malignant Biliary Obstruction | 53 | 50 | 103
  Biliary Stent Change | 25 | 25 | 50
  Biliary Leak | 11 | 12 | 23
  Increased Liver Tests/Jaundice | 13 | 9 | 22
  Pancreatic Stricture | 3 | 5 | 8
  Suspected Sphincter of Oddi Dysfunction (SOD) | 6 | 8 | 14
  Pancreatic Leak/Disruption | 11 | 12 | 23
  Pancreatic Duct Stone | 3 | 2 | 5
  Recurrent Acute Pancreatitis | 5 | 2 | 7
  Ampullectomy | 6 | 5 | 11
  Other | 16 | 31 | 47
History of post-ERCP Pancreatitis [Number; unit: participants]
  Yes | 9 | 9 | 18
  No | 214 | 217 | 431
History of Previous Sphincterotomy [Number; unit: participants]
  Yes | 72 | 71 | 143
  No | 151 | 155 | 306
Previous ERCP [Number; unit: participants]
  Yes | 81 | 79 | 160
  No | 142 | 147 | 289
Difficult Cannulation [Number; unit: participants] — Difficult Cannulation was defined by >8 attempts at cannulation
  participants
    Yes | 46 | 42 | 88
    No | 177 | 184 | 361
Precut Biliary Sphincterotomy [Number; unit: participants]
  Yes | 11 | 16 | 27
  No | 212 | 210 | 422
Therapeutic Biliary Sphincterotomy [Number; unit: participants]
  Yes | 106 | 114 | 220
  No | 117 | 112 | 229
Therapeutic Pancreatic Sphincterotomy [Number; unit: participants]
  Yes | 12 | 5 | 17
  No | 211 | 221 | 432
Minor Duct Sphincterotomy [Number; unit: participants]
  Yes | 5 | 4 | 9
  No | 218 | 222 | 440
Balloon Dilation of Biliary Sphincter [Number; unit: participants]
  Yes | 21 | 20 | 41
  No | 202 | 206 | 408
Wire Cannulation of Pancreatic Duct [Number; unit: participants]
  Yes | 90 | 89 | 179
  No | 133 | 137 | 270
Pancreatography [Number; unit: participants]
  Yes | 50 | 49 | 99
  No | 173 | 177 | 350
Pancreatic Acinarization [Number; unit: participants]
  Yes | 5 | 4 | 9
  No | 218 | 222 | 440
Biliary Strent Placement [Number; unit: participants]
  Yes | 89 | 84 | 173
  No | 134 | 142 | 276
Pancreatic Stent Placement [Number; unit: participants]
  Yes | 36 | 35 | 71
  No | 187 | 191 | 378
Trainee Involvement [Number; unit: participants]
  Yes | 152 | 168 | 320
  No | 71 | 58 | 129
Concomitant Endoscopic Ultrasound with Fine Needle Aspiration (EUS/FNA) [Number; unit: participants]
  Yes | 41 | 40 | 81
  No | 182 | 186 | 368
Periprocedural Fluid Volume [Mean (Standard Deviation); unit: Milliliters] | 705 (335) | 703 (355) | 704 (345)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Developed Acute Pancreatitis
Description: Number of patients who developed pancreatitis following ERCP based on Atlanta Classification
Time Frame: From randomization to 30 days after ERCP
Population: Patient who randomized into the study and received either rectal indomethacin or placebo
Measure: Number; unit: participants
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 223 | 226
participants | 16 | 11
Statistical Analysis 1: Comparison: Indomethacin vs Placebo; Test type: Superiority or Other; p = 0.33, Fisher Exact

2. Secondary Outcome: Number of Patients Who Developed Severe Pancreatitis
Description: Number of patients with severe acute pancreatitis based on the Atlanta Classification
Time Frame: From randomization to 30 days after ERCP
Population: Assess the number of patients who developed severe acute pancreatitis
Measure: Number; unit: participants
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 223 | 226
participants | 0 | 1
Statistical Analysis 1: Comparison: Indomethacin vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact

3. Secondary Outcome: Number of Patients Who Developed Moderately Severe Pancreatitis
Description: Number of patients with moderately severe pancreatitis based on Atlanta Classification
Time Frame: From randomization to 30 days after ERCP
Measure: Number; unit: participants
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 223 | 226
participants | 0 | 1
Statistical Analysis 1: Comparison: Indomethacin vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact

4. Secondary Outcome: Number of Patients Who Developed Mild Pancreatitis
Description: Number of patient who developed mild acute pancreatitis based on the Atlanta Classification
Time Frame: From randomization to 30 days after ERCP
Measure: Number; unit: participants
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 223 | 226
participants | 16 | 9
Statistical Analysis 1: Comparison: Indomethacin vs Placebo; Test type: Superiority or Other; p = 0.15, Fisher Exact

5. Secondary Outcome: Number of Patients Who Developed Gastrointestinal Bleeding
Description: Number of patients who developed any type of gastrointestinal bleeding from time of ERCP to 30 days post procedure
Time Frame: From randomization to 30 days after ERCP
Measure: Number; unit: participants
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 223 | 226
participants | 4 | 6
Statistical Analysis 1: Comparison: Indomethacin vs Placebo; Test type: Superiority or Other; p = 0.75, Fisher Exact

6. Secondary Outcome: Number of Patient Deaths
Description: Number of patients who died from any cause from the time of ERCP until 30 days post-procedure
Time Frame: From randomization to 30 days after ERCP
Measure: Number; unit: participants
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 223 | 226
participants | 0 | 3
Statistical Analysis 1: Comparison: Indomethacin vs Placebo; Test type: Superiority or Other; p = 0.25, Fisher Exact

7. Secondary Outcome: Number of Patients With 30 Days Hospital Re-admission
Description: Number of patients admitted to the hospital for any cause following ERCP
Time Frame: From randomization until 30 days after ERCP
Measure: Number; unit: participants
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 223 | 226
participants | 31 | 20
Statistical Analysis 1: Comparison: Indomethacin vs Placebo; Test type: Superiority or Other; p = 0.10, Fisher Exact

ADVERSE EVENTS:
Time Frame: From randomization to 30 days after ERCP
Arm/Group | Indomethacin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/223 | 3/226
Other Adverse Events (participants affected / at risk) | 4/223 | 6/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indomethacin (N=223) | Placebo (N=226)
Severe Acute Pancreatitis Leading to Death (Gastrointestinal disorders) | 0 (0) | 1 (1)
Secondary Bacterial Peritonitis due to Multifocal Hepatocellular Carcinoma Leading to Death (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aspiration Post-Procedure Leading to Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indomethacin (N=223) | Placebo (N=226)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 4 (4) | 6 (6) — Patients with any type of gastrointestinal bleeding

LIMITATIONS AND CAVEATS:
The study was terminated due to indomethacin's lack of efficacy after 449 patients had been enrolled. Thus the study may be underpowered to draw conclusions about the role of indomethacin in preventing post ERCP pancreatitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes